CLINICAL TRIAL: NCT00091377
Title: Multi-Center, Phase Ib/IIa Safety and Preliminary Efficacy Study of Phenoxodiol (Intravenous) as a Chemo-Sensitizing Agent for Cisplatin and Paclitaxel in Epithelial Ovarian Cancer or Primary Peritoneal Cancer, Platinum- and/or Taxane-Refractory or Resistant
Brief Title: Phenoxodiol Combined With Either Cisplatin or Paclitaxel in Patients With Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000389129; NOVOGEN-NV06-037; YALE-HIC-26423
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Paclitaxel; phenoxodiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Phenoxodiol IV 3 mg/kg combined with cisplatin 40 mg/m2 on Day 2 6 week cycles
  Interventions: Drug: cisplatin; Drug: phenoxodiol
- Arm B (Experimental): Phenoxodiol IV 3 mg/kg combined with paclitaxel 80 mg/m2 on Day 2 6 week cycles
  Interventions: Drug: paclitaxel; Drug: phenoxodiol

INTERVENTIONS:
Drug: cisplatin — IV 40 mg/m2 on Day 2 Number of Cycles: until progression or unacceptable toxicity or other withdrawal criteria are met.
  Arms: Arm A
Drug: paclitaxel — IV 80 mg/m2 on Day 2 Number of Cycles: until progression or unacceptable toxicity or other withdrawal criteria are met.
  Arms: Arm B
Drug: phenoxodiol — IV 3 mg/kg

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Phenoxodiol may help cisplatin and paclitaxel kill more tumor cells by making tumor cells more sensitive to the drugs.

PURPOSE: This randomized phase I/II trial is studying the side effects of phenoxodiol when given together with either cisplatin or paclitaxel and to see how well they work in treating patients with recurrent late-stage ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer that has not responded to treatment with drugs such as paclitaxel, docetaxel, cisplatin, or carboplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety and tolerability of phenoxodiol combined with cisplatin or paclitaxel in patients with recurrent late-stage ovarian epithelial, fallopian tube, or primary peritoneal cancer that is refractory or resistant to platinum and/or taxane drugs.
* Compare, preliminarily, tumor response in patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms according to medical history.

* Arm I: Patients receive phenoxodiol IV over 10 minutes on days 1 and 2 and cisplatin IV over 1 hour on day 2.
* Arm II: Patients receive phenoxodiol as in arm I and paclitaxel IV over 1 hour on day 2.

In both arms, treatment repeats every 6 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at 12, 24, 36, and 48 weeks or at the end of study participation.

Patients are followed at 6 and 12 months.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cancer

  * Recurrent disease
* Received no more than 4 prior chemotherapy regimens for this malignancy

  * Considered refractory or resistant to prior taxane (paclitaxel or docetaxel) and/or platinum (cisplatin or carboplatin) therapy based on 1 of the following criteria:

    * Treatment-free interval < 6 months after platinum or paclitaxel
    * Disease progression during platinum- or paclitaxel-based therapy
* Measurable or evaluable disease

  * Measurable disease is defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Evaluable disease is defined as doubling of CA 125 blood levels within the past 6 months AND CA 125 level ≥ 2 times upper limit of normal (ULN) within the past week
* No active CNS metastases

  * Patients with known CNS metastases must have received prior radiotherapy or CNS-directed chemotherapy AND have ≥ 4 weeks of stable disease

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* Hematocrit ≥ 28% (transfusion or growth factors allowed)
* Hemoglobin > 8.0 g/dL (transfusion or growth factors allowed)

Hepatic

* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No neuropathy (sensory or motor) > grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy for the malignancy

Radiotherapy

* See Disease Characteristics
* No prior whole abdominal radiotherapy
* Concurrent localized radiotherapy allowed for control of local complications not indicative of general disease progression

Surgery

* Not specified

Other

* Recovered from prior antineoplastic therapy
* More than 4 weeks since prior standard therapy for malignant tumor
* More than 6 months since prior investigational anticancer drugs
* No other concurrent investigational drugs
* No concurrent drugs significantly metabolized by the cytochrome P450 enzymes CYP2C8, CYP2C9, CYP2C19, and CYP3A4/B1C
* No concurrent amifostine or other protective agents
* No concurrent grapefruit juice

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Average 6 mo
Efficacy | Average 6 months

SECONDARY OUTCOMES:
Surrogate marker of tumor response in terms of plasma protein tNOX | Average 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren Lancaster, Study Chair — Kazia Therapeutics Limited
Locations (2):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States
- Royal Women's Hospital, Carlton, Victoria, Australia

REFERENCES:
- [Result] Kelly MG, Mor G, Husband A, O'Malley DM, Baker L, Azodi M, Schwartz PE, Rutherford TJ. Phase II evaluation of phenoxodiol in combination with cisplatin or paclitaxel in women with platinum/taxane-refractory/resistant epithelial ovarian, fallopian tube, or primary peritoneal cancers. Int J Gynecol Cancer. 2011 May;21(4):633-9. doi: 10.1097/IGC.0b013e3182126f05. PMID 21412168